CLINICAL TRIAL: NCT05990530
Title: Evaluation of the Efficacy and Safety of Allogeneic Transplantation of Expanded Pancreatic Islet Cells in Patients With "Brittle" Type 1 Diabetes
Brief Title: Allogeneic Transplantation of Expanded Pancreatic Islet Cells
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YD02-2022
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Brittle Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YD02-2022 (Experimental)
  Interventions: Biological: YD02-2022

INTERVENTIONS:
Biological: YD02-2022 — Human islet cells were isolated and expanded in vitro to generate islets containing all types of pancreatic endocrine cells and possessing comparable function of human islets. These islet cells will be infused into the hepatic portal vein.

SUMMARY:
This study will evaluate the efficacy and safety of allogeneic pancreatic islet cells transplantation in patients with "brittle" type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form and agree to comply with the trial treatment plan and visit schedule.
2. Age ≥18 years and ≤60 years on the day of signing the informed consent form, regardless of gender.
3. Body mass index (BMI) ≥18.0 kg/m2 and ≤35.0 kg/m2.
4. Diagnosed with T1DM based on the World Health Organization's diabetes classification (2019).
5. HbA1c ≥7.0% and ≤15.0% at screening.
6. Dependence on insulin injection therapy for ≥5 years, receiving a stable insulin treatment plan for ≥3 months, and injecting insulin three or more times per day or using an insulin pump.
7. Postprandial mixed meal stimulated C-peptide level <0.3 ng/mL.
8. Experienced impaired awareness of hypoglycemia or significant glycemic instability during screening and in the past 6 months. Hypoglycemic episodes are associated with impaired awareness of hypoglycemia, extreme glycemic instability, or severe fear and maladaptive behavior.
9. Sexually active males who are not surgically sterilized or have partners of childbearing potential agree to use effective contraception during the entire trial period and for at least 6 months after the study ends; sexually active females of childbearing potential agree to use effective contraception during the entire study period and for at least 6 months after the study ends.

Exclusion Criteria:

1. Types of diabetes other than T1DM.
2. Body mass index (BMI) >35 kg/m2 or weight <50 kg.
3. Excessive insulin sensitivity and/or insulin resistance (insulin requirement >1.0 IU/kg/day or <15 U/day).
4. Previous pancreatic or islet transplantation. Severe trauma, severe infection, or surgery that may affect glycemic control within one month before screening.
5. History of hypertension with systolic blood pressure (SBP) >160 mmHg and/or diastolic blood pressure (DBP) >100 mmHg after stable dose (at least 4 weeks) of antihypertensive medication.
6. Blood transfusion or severe bleeding within the past 3 months, known hemoglobin-related diseases, anemia (moderate to severe), or other known hemoglobinopathies that interfere with HbA1c measurement (such as sickle cell disease).
7. Impaired liver or kidney function at screening: aspartate aminotransferase (AST) ≥3 times the upper limit of normal (ULN), alanine aminotransferase (ALT) ≥3 times ULN, total bilirubin level (TBL) ≥2 times ULN (excluding Gilbert's syndrome), creatinine clearance rate <45 mL/min (calculated by the Cockcroft-Gault formula).
8. Significant albuminuria (urinary albumin excretion rate >300 mg/g) or history thereof.
9. Uncontrolled or untreated thyroid disease or adrenal insufficiency.
10. Severe diabetic kidney disease or renal insufficiency, proliferative retinopathy, diabetic foot ulcers, diabetes-related amputation, and/or severe peripheral neuropathy at screening.
11. Active hepatitis B, hepatitis C, acquired immunodeficiency syndrome, syphilis, or tuberculosis. Even without clinical evidence of active infection, participants with laboratory evidence of active infection are also excluded.
12. Severe heart disease or a history of cardiovascular disease within 6 months before screening, including stroke, decompensated heart failure (NYHA class III or IV), myocardial infarction, unstable angina, or coronary artery bypass grafting.
13. Previous history of coagulation disorders or requiring long-term anticoagulant therapy (e.g., warfarin) (low-dose aspirin therapy is allowed) or patients with INR >1.5.
14. Substance abusers with a history of drug abuse/dependence or drug use within 1 year before screening.
15. Received live vaccines within 14 days before screening or planned to receive live vaccines during the trial or within 1 month after treatment. Live vaccines include, but are not limited to, measles, mumps, rubella, varicella, yellow fever, rabies, Bacillus Calmette-Guérin, typhoid vaccine, COVID-19 vaccine, etc.
16. Patients with a history of acute or chronic pancreatitis, symptomatic gallbladder disease, pancreatic injury, or other high-risk factors for pancreatitis, or patients with blood amylase >1.2 times ULN at screening.
17. Other abnormal laboratory test results deemed clinically significant by the investigator.
18. Patients with severe mental illness.
19. Participated in a drug or medical device clinical trial within the past 3 months and received investigational drugs or medical devices; or within 5 half-lives of another drug before screening (if the half-life exceeds 3 months).
20. Currently receiving long-term (continuous for ≥14 days) systemic pharmacological doses of glucocorticoids or other medications that may affect the participant's consciousness.
21. Treatment (local, intra-articular, intraocular, or inhalation preparations) for any other factors or diseases not mentioned above, deemed unsuitable for participation in this clinical study by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Residual β-Cell function (RBCF) | 12 months post-transplant
  Evaluation of the magnitude of C-peptide change after transplantation

SECONDARY OUTCOMES:
Glycemic control (HbA1c) | 52 weeks post-transplant
  Evaluation of the proportion of subjects with HbA1c ≤7.0% and no severe hypoglycemic events
Treatment (insulin-independent) | 12 weeks and 52 weeks post-transplant
  Evaluation of the proportion of subjects who are insulin-independent
Treatment (insulin requirement) | 12 weeks and 52 weeks post-transplant
  Evaluation of the percentage reduction in insulin requirement
Glycemic control (MAGE) | 12 weeks and 52 weeks post-transplant
  Evaluation of the average amplitude of glycemic fluctuations (MAGE) in subjects
Hypoglycemia (HYPO) | baseline and 52 weeks post-transplant
  Evaluation of the severity of hypoglycemia using the Ryan Hypoglycemia Severity Score (HYPO)
Quality of life score | baseline and 52 weeks post-transplant
  Evaluation of the quality of life score in subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology and Metabolic Diseases, Ruijin Hospital, Shanghai Jiao-Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided